CLINICAL TRIAL: NCT06649084
Title: Establishing Evidence-based Multicomponent Treatment for Speech and Language in Primary Progressive Aphasia
Brief Title: Primary Progressive Aphasia Multicomponent Language Treatment Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Maya Henry, Associate Professor, University of Texas at Austin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R56DC016291 (NIH); R56DC016291 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Primary Progressive Aphasia; Semantic Dementia; Semantic Memory Disorder; Logopenic Progressive Aphasia; Nonfluent Aphasia, Progressive; Aphasia; Aphasia, Progressive
Keywords: Speech-Language Pathology; Neurodegenerative Disease; Logopenic; Semantic; Nonfluent; Speech Entrainment; Telethearpy; Multimodal Communication Training; Partner Training; Augmentative and Alternative Communication; Script training
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia; Memory Disorders; Primary Progressive Nonfluent Aphasia; Aphasia; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Multicomponent Lexical Retrieval Training (Multi-LRT) (Experimental)
  Interventions: Behavioral: Multicomponent Lexical Retrieval Training (Multi-LRT)
- Multicomponent Video Implemented Script Training in Aphasia (Multi-VISTA) (Experimental)
  Interventions: Behavioral: Multicomponent Video Implemented Script Training in Aphasia (Multi-VISTA)
- Experimental: Multicomponent Communicaiton Partner Training (Multi-CPT) (Experimental)
  Interventions: Behavioral: Multicomponent Communication Partner Training (Multi-CPT)

INTERVENTIONS:
Behavioral: Multicomponent Lexical Retrieval Training (Multi-LRT) — In person or via teletherapy: A multi-component treatment incorporating elements of restitutive, compensatory, and care-partner focused interventions. Participants work on producing names of personally relevant target in multiple communication modalities. Treatment focuses on the use of strategies which capitalize on residual linguistic ability and autobiographical memory to support word retrieval. The participant completes two one-hour-long sessions per week plus daily homework. The participant also meets 4 times during the course of treatment with a study partner (e.g., spouse) for communication counseling, education, and practice of communication strategies.
  Arms: Multicomponent Lexical Retrieval Training (Multi-LRT)
Behavioral: Multicomponent Video Implemented Script Training in Aphasia (Multi-VISTA) — In person or via teletherapy: A multi-component treatment incorporating elements of restitutive, compensatory, and care-partner focused interventions. Participants work on producing personally relevant scripts of 3-5 sentences in length. Length and complexity of scripts are individually tailored. The participant completes 30 minutes per day of home practice, during which they speak in unison with a video/audio model of a healthy speaker clearly articulating the scripts. Biweekly (one hour each) sessions with a clinician are held which target clear and accurate script production, script memorization, and conversational usage of the script and multimodal communication. The participant also meets 6 times during the course of treatment with a study partner (e.g., spouse) for communication counseling, education, and practice of communication strategies.
  Arms: Multicomponent Video Implemented Script Training in Aphasia (Multi-VISTA)
Behavioral: Multicomponent Communication Partner Training (Multi-CPT) — In person or via teletherapy: A multi-component treatment incorporating elements of compensatory and care-partner focused interventions. Biweekly (one hour each) sessions with a clinician are held which target use of communication strategies including multimodal communication for the participant and study partner (e.g., spouse). The participant also completes regular assignments meant to increase generalization of communication strategies and progress on personal goals.
  Arms: Experimental: Multicomponent Communicaiton Partner Training (Multi-CPT)

SUMMARY:
The goal of this clinical trial is to learn if a speech-language telerehabilitation helps improve communication in people with primary progressive aphasia (PPA), a form of dementia that affects speech and language. The study will also document how acceptable and helpful the program is for both patients and their care partners.

The main questions the study aims to answer are:

1. Is the telerehabilitation program feasible and acceptable for people with PPA and their care partners?
2. Do participants with PPA and care partners report satisfaction with the program?
3. Which outcome measures are most useful for evaluating changes in communication and quality of life?
4. What patterns of treatment response are seen in participants after completing the program?

Researchers will test the program in a small group of participants to see how people respond. The program includes both speech-language therapy and training for care partners.

Participants will:

* Take part in online speech-language therapy sessions
* Complete communication tasks and questionnaires before and after the program
* Have regular virtual check-ins with the research team
* Include their care partners in some parts of the program for training and support

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for Primary Progressive Aphasia (PPA; Gorno-Tempini et al., 2011)
* Scores of 10 or higher on the Mini-Mental State Examination
* Has a study partner who can consistently attend sessions

Exclusion Criteria:

* Other neurological or psychiatric diagnosis that may contribute to cognitive-linguistic deficits
* Significant, uncorrected visual or hearing impairment that would interfere with participation
* Score of less than 10 on the Mini-Mental State Examination
* Prominent initial non-speech-language impairment (cognitive, behavioral, motoric)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in script production accuracy | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment
  Percent correct intelligible, scripted words for trained/untrained scripts
Change in spoken naming of trained/untrained items | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment
  Percent correctly named trained/untrained pictures
Information communicated in any modality for trained/untrained stimuli | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment
  Percent of major content units (key words) communicated via speech or nonspeech modalities (e.g., writing, drawing, gesture) for trained/untrained scripts (Multi-VISTA) or words (Multi-LRT) during structured probes and in conversation
Goal Attainment Score | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment
  The Goal Attainment Score is self-reported progress on personalized goals based on a five point scale.

SECONDARY OUTCOMES:
Change on Quick Aphasia Battery | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment
  change on standardized aphasia assessment
Change on Aphasia Impact Questionnaire | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment
  change on psychosocial questionnaire for individuals with aphasia

OTHER OUTCOMES:
Post-treatment Communication Survey | post-treatment (approximately 6-12 weeks after treatment onset)
  survey characterizing perceived response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maya L Henry, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No